CLINICAL TRIAL: NCT01788085
Title: RD-41 Development of Applications of the Bravo® pH Monitoring System and Evaluation of Its Performance
Brief Title: Development of Applications of the Bravo® pH Monitoring System and Evaluation of Its Performance (Encore)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-41
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Gastro Esophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pH monitoring procedure (Experimental): Bravo pH monitoring procedure
  Interventions: Device: Bravo pH monitoring procedure

INTERVENTIONS:
Device: Bravo pH monitoring procedure — Bravo pH monitoring procedure

SUMMARY:
Study Hypothesis: This study is designed as an integral part of the development of new or improved features or components of the Bravo® pH Monitoring System and may serve verification and validation purposes.

The study population will include symptomatic patients with known or suspected gastroesophageal reflux disease

Symptomatic patients will undergo invasive procedure, including Bravo capsule delivery, positioning and attachment. Confirmation of capsule attachment may be done endoscopically.

These procedures will serve to evaluate overall system performance in actual clinical setup, for instance: ergonomics and performance of delivery device, capsule transmission etc.

Physician may be asked to provide feedback on the procedure and/or document their activities during the procedure.

DETAILED DESCRIPTION:
The study population consists of symptomatic patients with known or suspected gastro esophageal reflux disease. The aim of this clinical study is to evaluate Bravo® pH Monitoring System.

Primary objectives

* To evaluate usability and functionality of the Bravo® pH Monitoring System and procedure
* To evaluate modifications to the Bravo delivery device Primary Endpoints

  1. Evaluate physician subjective assessment questionnaire (appendix 3)
  2. Percentage of successful capsule attachments Patients will undergo standard-of-care Bravo pH procedure. Prior to the pH study, the patient should not eat or drink for a minimum of 6 hours, according to the standard system instructions.
* Bravo procedure may take 48-96 hours
* Patients will have a follow-up visit or call, one to two weeks after the procedure
* A fluoroscopy procedure may be ordered at physician's discretion to verify capsule attachment \ detachment from the patient's esophagus

Over all expected duration for subject's participation in the study will be a maximum of 1 month

Physician may be asked to provide feedback on the procedure usability and functionality and to document their activities during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 years old
2. Subject received an explanation about the nature of the study and agrees to provide written informed consent.
3. The subject was referred for pH monitoring procedure to detect acid reflux for at least one of the following reasons:

   * Burning substernal chest pain (heartburn)
   * Regurgitation of food or stomach contents
   * Dysphagia
   * Epigastric pain
   * Non-erosive reflux disease (NERD)
   * Chest pain
   * Cough
   * Hoarseness
   * Asthma
   * Lower pharyngeal irritation, need to clear throat

Exclusion Criteria:

1. Subject has a cardiac pacemaker or other implanted electromedical device.
2. Subject has any condition, which precludes compliance with study and/or device instructions.
3. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
4. Subject suffers from life threatening conditions
5. Subject currently participating in another clinical study which may interfere with study objectives, per physician discretion
6. Subject has prior abdominal surgery other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
7. Subject is schedule to undergo MRI examination within 30 days from pH monitoring procedure.
8. Subject has known bleeding diathesis, strictures, severe esophagitis, varices and or obstructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate physician subjective assessment questionnaire | post Bravo pH monitoring pinning procedure, same day of procedure
Percentage of successful capsule attachments | post Bravo pH monitoring pinning procedure, same day of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lavy, Prof., Principal Investigator — Bnei Zion MC, HAifa, Israel
Locations (1):
- Bnei-Zion MC, Haifa, Israel